CLINICAL TRIAL: NCT05388175
Title: Time of Device Positioning of LISA Rigid Catheter vs LISA Soft Catheter in a Very Preterm Manikin: A Crossover Randomized Controlled Trial
Brief Title: LISA Rigid Catheter vs LISA Soft Catheter in a Very Preterm Manikin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Associate Professor, University Hospital Padova
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NEOUNIPD1(2022)
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Respiratory Distress Syndrome in Preterm Infants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician will be blinded of the treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Less invasive surfactant administration (LISA) with a rigid catheter (Experimental): Participants will simulate the procedure of surfactant administration by using a rigid catheter
  Interventions: Device: Rigid catheter
- Less invasive surfactant administration (LISA) with a soft catheter (Active Comparator): Participants will simulate the procedure of surfactant administration by using a soft catheter
  Interventions: Device: Soft catheter

INTERVENTIONS:
Device: Rigid catheter — Participants will be invited to positioning a rigid catheter in the manikin's trachea for surfactant aministration
  Other Names: Less invasive surfactant administration (LISA) with a rigid catheter
  Arms: Less invasive surfactant administration (LISA) with a rigid catheter
Device: Soft catheter — Participants will be invited to positioning a rigid catheter in the manikin's trachea for surfactant aministration
  Other Names: Less invasive surfactant administration (LISA) with a soft catheter
  Arms: Less invasive surfactant administration (LISA) with a soft catheter

SUMMARY:
Less invasive surfactant administration (LISA) can be provided using rigid or soft catheters, but possible differences in terms of easiness of use and success of the procedure are unknown. A difficult procedure may have some drawbacks such as the prolonged duration of the laryngoscopy needed to insert the device, which is likely to aggravate the invasiveness of the procedure and result in stressful consequences such as bradycardia, hypoxia, and hemodynamic changes.

Objectives: i) time of device positioning, ii) success of the procedure of positioning the device, iii) participant's satisfaction.

DETAILED DESCRIPTION:
This is an unblinded, randomized, controlled, crossover (AB/BA) trial of surfactant treatment with LISA with a rigid catheter vs. LISA with a soft catheter in a manikin simulating an extremely low birth weight infant. Participants will be level III NICU consultants and residents. Randomization will be performed using a computer-generated random assignment list. The primary outcome measure will be the total time of device positioning. The secondary outcomes will be the success of the first attempt, the number of attempts to achieve the correct positioning of the device in the trachea, the achievement of the correct depth of the catheter in the trachea, and the participant's opinion on using the device.

ELIGIBILITY:
Inclusion Criteria:

* Level III NICU consultants and residents will be eligible to participate in the study

Exclusion Criteria:

* There are no exclusion criteria for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Total time of device (catheter) positioning | 5 minutes
  The time of device positioning defined as the time elapsed from the positioning of the laryngoscope in the manikin mouth to the connection of the syringe for surfactant administration to the catheter

SECONDARY OUTCOMES:
Success of device positioning at the first attempt | 1 minute
  We will evaluate the success of the device (catheter) at the first attempt
Achievement of the correct depth of the catheter in the trachea | 5 minutes
  The correct depth of the catheter tip in the trachea will be evaluated by an external observer
Participant's opinion regarding the procedure | 5 minutes
  Participant's opinion regarding the feasibility or difficulty of the procedure will be evaluated by using a questionnaire with items (1 worse to 5 best outcome) to be evaluated by a Likert scale

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Poliambulanza Breacia, Brescia
  - Azienda Ospedaliera di Padova, University of Padova, Padua

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared upon motivated request to the PI
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: Upon motivated request to the PI